CLINICAL TRIAL: NCT03995589
Title: Exercise Therapy in Patients With Peripheral Artery Disease: Evaluating the Clinical Effectiveness of Exercise Therapy and Exploring Determinants of Improvement
Acronym: PROSECO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Véronique Cornelissen, Assistant Professor, KU Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s9acq68z
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking Group (Experimental)
  Interventions: Other: Walking
- Control (Active Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Other: Walking — Technology-guided semi-supervised walking therapy
  Arms: Walking Group
Other: Control — Go Home and Walk advice
  Arms: Control

SUMMARY:
I. To investigate whether patient characteristics, exercise therapy characteristics, local metabolic exercise response, endothelial function, autonomic function or atherosclerotic lesion location can predict the walking response to a successfully completed semi-supervised exercise intervention in patients with intermittent claudication (WP I) II. To assess the effect of a home-based exercise intervention with remote monitoring and coaching on cardiovascular risk factors in patients with intermittent claudication (WP II)

ELIGIBILITY:
The study population will comprise patients diagnosed with lower-extremity artery disease (ABI ≤0.9 and/or 20% decrease after a maximal treadmill test) suffering from intermittent claudication (Rutherford 1-3) presenting with new complaints (at least 6 months after previous revascularization) at the Vascular Center of university hospitals Leuven will be included if according to current guidelines their initial treatment should be conservative

Inclusion Criteria:

* age > 17 yrs
* ABI ≤0.9 and/or 20% decrease after a maximal treadmill test
* intermittent claudication (Rutherford 1-3)
* ability to undertake an exercise test and read and understand Dutch questionnaires

Exclusion criteria

* exercise test induced signs of complex arrhythmias or significant ischemia during baseline testing
* other comorbidity limiting participation in the exercise group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Pain free walking distance | Baseline - 12 weeks
  Treadmill protocol

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cornelis N, Buys R, Fourneau I, Van den Bosch A, De Wilde C, Goetschalckx K, Cornelissen V. Cardiorespiratory fitness in patients with lower extremity artery disease? It takes more than just some steps! Eur J Prev Cardiol. 2022 May 5;29(5):e190-e192. doi: 10.1093/eurjpc/zwab135. No abstract available. PMID 34417620